CLINICAL TRIAL: NCT01375829
Title: Phase I Study of Ixabepilone and Temsirolimus in Adult Patients With Advanced Solid Tumors
Brief Title: Ixabepilone and Temsirolimus in Treating Patients With Solid Tumors That Are Metastatic or Cannot Be Removed by Surgery
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02907; NCI-2012-02907 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-2012-01136; CDR0000702380; NCI-2011-01140; MC1013 (Other: Mayo Clinic in Rochester); 8814 (Other: CTEP); P30CA015083 (NIH); U01CA069912 (NIH); UM1CA186686 (NIH); NCT02344147 (obsolete NCT alias)
Record Dates: First submitted 2011-06-16; First posted 2011-06-17 (Estimated); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Adult Solid Neoplasm
MeSH Terms: interventions — ixabepilone; Epothilones; temsirolimus; Sirolimus

ARMS (1):
- Treatment (ixabepilone, temsirolimus) (Experimental): Patients receive ixabepilone IV over 3 hours on day 1 and temsirolimus IV over 30-60 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ixabepilone; Other: Pharmacological Study; Drug: Temsirolimus

INTERVENTIONS:
Drug: Ixabepilone — Given IV
  Other Names: (1S,3S,7S,10R,11S,12S,16R)-7,11-Dihydroxy-8,8,10,12,16-pentamethyl-3-[(1E)-1-methyl-2-(2-methyl-4-thiazolyl)ethenyl]-17-oxa-4-azabicyclo[14.1.0]heptadecane-5,9-dione; Azaepothilone B; BMS 247550; BMS-247550; BMS247550; Epothilone; Epothilone-B BMS 247550; Ixempra
Other: Pharmacological Study — Correlative studies
Drug: Temsirolimus — Given IV
  Other Names: CCI 779; CCI-779; CCI-779 Rapamycin Analog; CCI779; Cell Cycle Inhibitor 779; Rapamycin Analog; Rapamycin Analog CCI-779; Torisel

SUMMARY:
This phase I trial studies the side effects and best dose of ixabepilone and temsirolimus in treating patients with solid tumors that have spread from the primary site to other places in the body or cannot be removed by surgery. Drugs used in chemotherapy, such as ixabepilone, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Temsirolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving ixabepilone together with temsirolimus may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximally tolerated dose (MTD) of the combination of ixabepilone and temsirolimus in patients with advanced solid tumors.

II. To describe toxicity profiles associated with the combination of ixabepilone and temsirolimus.

III. To assess preliminary efficacy of the combination of ixabepilone and temsirolimus.

OUTLINE: This is a dose-escalation study.

Patients receive ixabepilone intravenously (IV) over 3 hours on day 1 and temsirolimus IV over 30-60 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with histologically confirmed solid tumor malignancy that is metastatic or unresectable and for which standard curative measures or other therapy that provide survival benefit do not exist or are no longer effective
* Patients may not have had more than two systemic therapeutic regimens in the metastatic disease setting with the following exceptions: hormonal therapy (e.g. tamoxifen, aromatase inhibitors, anti-androgen therapy, etc.)
* Patients with non-measurable, but assessable, disease will be allowed
* Absolute neutrophil count >= 1500/mcL
* Hemoglobin >= 9.0 g/dL
* Platelets >= 100,000/mcL
* Total bilirubin < 1.5 mg/dL
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) or serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) =< 2.5 x institutional upper limit of normal (ULN) in the absence of hepatic metastasis; SGPT (ALT) =< 3 x ULN or SGOT (AST) =< 5 x ULN in the presence of hepatic metastasis
* Creatinine =< 1.5 x ULN
* International normalized ratio (INR) =< 1.4 for patients not on warfarin (Coumadin)
* INR range of 2.0-3.0 for patients on therapeutic doses of warfarin (Coumadin)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2
* Ability to provide informed consent
* Willingness to return to a Mayo Clinic institution for follow up
* Life expectancy >= 84 days (12 weeks)
* Women of childbearing potential only: negative serum pregnancy test done =< 7 days prior to registration

Exclusion Criteria:

* Known standard therapy for the patient's disease that is potentially curative or definitely capable of extending life expectancy
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, uncontrolled diabetes or with hemoglobin A1c (HbA1C) > 8, or psychiatric illness/social situations that would limit compliance with study requirements
* Any of the following prior therapies:

  * Chemotherapy =< 28 days prior to registration
  * Mitomycin C/nitrosoureas =< 42 days prior to registration
  * Immunotherapy =< 28 days prior to registration
  * Biologic therapy =< 28 days prior to registration
  * Radiation therapy =< 28 days prior to registration
  * Radiation to > 25% of bone marrow
* Failure to fully recover from acute, reversible effects of prior chemotherapy regardless of interval since last treatment
* New York Heart Association classification III or IV
* Known central nervous system (CNS) metastases or seizure disorder; patients with known brain metastases that have been successfully treated and stable for > 6 months without requirement for corticosteroids and without seizure activity will be eligible
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational (utilized for a non-Food and Drug Administration [FDA]-approved indication and in the context of a research investigation)
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients (other than that related to the use of corticosteroids) including patients known to be human immunodeficiency virus (HIV) positive
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* History of myocardial infarction =< 168 days (6 months), or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* >= Grade 2 sensory neuropathy
* >= Grade 2 hypertriglyceridemia
* >= Grade 2 hypercholesterolemia
* Patients on medication considered strong cytochrome P450 3A4 (CYP3A4) inducers (efavirenz, nevirapine, carbamazepine, phenobarbital, phenytoin, pioglitazone, rifabutin, rifampin, St. John's wort) or CYP3A4 inhibitors (indinavir, nelfinavir, ritonavir, clarithromycin, itraconazole, ketoconazole, nefazodone, saquinavir, telithromycin) unless the medication can be substituted with another agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-06-27 (Actual); Primary Completion 2018-06-26 (Actual); Study Completion 2026-03-19 (Estimated)

PRIMARY OUTCOMES:
MTD of the combination of ixabepilone and temsirolimus, defined as the dose level below the lowest dose that induces dose-limiting toxicity in at least one-third of patients (at least 2 of a maximum of 6 new patients) | 21 days

SECONDARY OUTCOMES:
Incidence of adverse events graded according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | Up to 3 months
  The number and severity of all adverse events (overall, by dose-level, and by tumor group) will be tabulated and summarized in this patient population.
Incidence of overall toxicity graded according to Common Toxicity Criteria standard grading | Up to 3 months
  Frequency distributions, graphical techniques and other descriptive measures will form the basis of these analyses.
Best response, defined to be the best objective status recorded from the start of the treatment until disease progression/recurrence | Up to 3 months
  Responses will be summarized by simple descriptive summary statistics delineating complete and partial responses as well as stable and progressive disease in this patient population (overall and by tumor group).
Time until any treatment related toxicity | Up to 3 months
Time until treatment related grade 3+ toxicity | Up to 3 months
Time until hematologic nadirs (white blood cells, absolute neutrophil count, platelets) | Up to 3 months
Time to progression | Up to 3 months
Time to treatment failure | From registration to documentation of progression, unacceptable toxicity, or refusal to continue participation by the patient, assessed up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Keith C Bible, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota